CLINICAL TRIAL: NCT01086020
Title: Same Lipid Lowering by Atorvastatin Versus Atorvastatin Plus Ezetimibe on Coronary Plaque Progression
Brief Title: Atorvastatin Plus Ezetimibe on Coronary Plaque Progression
Acronym: AEPP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Weifeng Shen, ruijin hospital, shanghai jiao tong university school of medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH20100101
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
Keywords: IVUS; coronary plaque; regression
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin; Ezetimibe

ARMS (2):
- atorvastatin (Active Comparator): patients will be treated with atorvastatin 10mg/d after randomization, and continued for two years
  Interventions: Drug: atorvastatin
- atorvastatin and ezetimibe (Experimental): patients will be treated with atorvastatin 5mg/d and Ezetimibe 5mg/d after randomization, and continued for two years
  Interventions: Drug: atorvastatin plus ezetimibe

INTERVENTIONS:
Drug: atorvastatin — Patients admitted with 20-70% coronary artery plaque identified by angiography will be treated with atorvastatin 10mg/d for two years
  Other Names: Lipitor
  Arms: atorvastatin
Drug: atorvastatin plus ezetimibe — Patients admitted with 20-70% coronary artery plaque identified by angiography will be treated with atorvastatin 5mg/d and Ezetimibe 5mg/d for two years
  Other Names: Lipitor and ezetrol
  Arms: atorvastatin and ezetimibe

SUMMARY:
Atherosclerosis is a progressive disease. Lipid lowering therapy was the standard treatment for patients with coronary artery disease. Studies indicated that coronary artery plaque progression had positive relationship with the plasma cholesterol level, and could be halted or reversed by intensive statin therapy (such as 20-40 mg/d atorvastatin). Ezetimibe plus statin could further lowered blood cholesterol level. Here the investigators hypothesize that same cholesterol lowering level by routing dose of atorvastatin or lower dose of atorvastatin plus ezetimibe could achieve the same effect on coronary artery plaque cessation or regression.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive the coronary angiography and potential PCI therapy

Exclusion Criteria:

* Patients was treated by statins before randomization
* Patient with ≤ 20% and ≥ 70% coronary narrowing and target lesion
* ST elevation myocardial infarction less than 7 days
* Without informed consent
* Abnormal liver function before randomization, (AST, ALT ≥ULN)
* Active hepatitis or muscular disease
* Impaired renal function with serum creatinine level > 3mg/dl
* Impaired left ventricular function with LVEF > 30%
* Participate in other studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
change of coronary artery plaque volume | 1 year
  The primary endpoint was the change of coronary artery plaque volume measured by intravascular ultrasound (IVUS) at one year after randomization.

SECONDARY OUTCOMES:
composite of adverse cardiac events | 2 years
  The secondary endpoint was the composite of adverse cardiac events (MACE), including cardiac death, non-fatal infarction and target vessel revascularization at two years after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Shen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital,, Shanghai, Shanghai Municipality, China